CLINICAL TRIAL: NCT00783029
Title: Reproducibility of Dynamic Vessel Analyzer Measurements and Establishment of Standards
Brief Title: Measurement of the Eye's Blood Vessels Using the Dynamic Vessel Analyzer (DVA)
Status: Completed | Type: Observational
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, Kerstin Bettermann, MD, PhD, Penn State University
Other Study IDs: HMC29113; IRB # 29113
Record Dates: First submitted 2008-10-30; First posted 2008-10-31 (Estimated); Last update posted 2012-02-07 (Estimated); Status verified 2012-02

CONDITIONS: Healthy
Keywords: Vasodilation; Vessel Reactivity; Dynamic Vessel Analyzer; Retina
MeSH Terms: conditions — Aneurysm

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy Subjects: Healthy participants between the ages of 21 and 65 years old.

SUMMARY:
The purpose of this research study is examine the response of the blood vessels in the eye to a light flicker stimulus using the Dynamic Vessel Analyzer (DVA) on two separate days in healthy individuals. The DVA uses an instrument which is used during routine eye examinations. The hypothesis of the study is that the changes in eye's blood vessel will be similar between the two visits; thus establishing reproducibility of the measurements for future comparisons to individuals with stroke or heart disease. In addition, this study will compare the eye's blood vessel responses to responses of the blood vessels in the arm using Doppler ultrasound.

DETAILED DESCRIPTION:
Retinal blood vessels have been suggested to be an index of the cerebral and coronary microvasculature function. Since the retinal vessels are not under direct sympathetic control, this vascular bed is an ideal location to examine local mechanisms of vascular regulation(i.e. metabolite/endothelial and myogenic). Based on previously published data on animal and human responses, the central purpose for the proposed research is to compare the retinal and brachial vasodilatation responses in healthy subjects using the Dynamic Vessel Analyzer (DVA). Our rationale for this proposal is to better understand retinal blood flow in healthy individuals, gain insight into vascular reactivity in different vascular beds, and lastly to establish standards and reproducibility of DVA Measurements.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Individuals
* Age: 21 to 65 years
* Non-smokers
* Non-obese

Exclusion Criteria:

* History of cardiovascular, pulmonary, peripheral vascular disease, renal, prostate, and urinary retention disease; Hypertension; Narrow angle Glaucoma or Age Related Macular Degeneration.
* Pregnancy
* Inability to fixate using eye device
* Does not wish to participate

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Subjects
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2008-10; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
To characterize changes in the diameter of retinal blood vessels to a light-induced flicker stimulus in healthy subjects on two separate visits. | 1 Year

SECONDARY OUTCOMES:
To compare retinal vasodilator responses to brachial reactive hyperemic responses. | 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: Kerstin Bettermann, MD, PhD, Principal Investigator — Penn State College of Medicine
Locations (1):
- Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States